CLINICAL TRIAL: NCT02646293
Title: Nephron Sparing Renal Surgery and Total Nephrectomy - Functional Adaptation, Preservation and Prediction of Kidney Function
Brief Title: Nephron Sparing Renal Surgery and Total Nephrectomy
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, Urologist, Zealand University Hospital
Other Study IDs: SN-43-2012
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of the diagnosis of renal cell carcinoma has increased during the past two decades because of the detection of small renal tumours that occur incidentally because of increased use of CT-scanning (1,2). Postoperative renal insufficiency was a significant independent predictor of overall and cardiovascular specific survival (3). "Nephron-sparing" surgical techniques are now preferred for small tumor masses and laparoscopic intervention is replacing open surgery at centers that master this technique. This is an area of priority within the Regions of Zaeland and Southern Denmark.

The primary endpoint is:

The early plasma (5 days) [NT-proBNP] response predicts long-term total renal function and function of the remaining kidney.

The second endpoint:

Plasma [NT-proBNP] increases acutely after partial nephrectomy and the change reflects the renal mass reduction.

Chronic blood pressure change is inversely related to plasma [BNP].

DETAILED DESCRIPTION:
Irreversible kidney damage is described beyond thirty minutes of warm ischemia time (WIT), even in completely normal systems (4). Gill et al. (5) reported 18% kidney function loss after thirty-two minutes of WIT. Preliminary data from our center shows a reduction in WIT to eleven minutes (6) associated with a reduction in renal function loss to 11%. There is however, an increasing need to understand the pathophysiology associated with partial nephrectomy procedure beyond the ischemia time and a need for biomarkers with predictive value in order to create an evidence-based, mechanistic frame for protective intervention. The current proposal seeks to address these issues in this highly specialized area.

Specific background for the study After unilateral total nephrectomy, the contralateral kidney within hours undergoes a functional adaptation with an increase in renal blood flow (RBF) and glomerular filtration rate(GFR) and thereby maintains whole body fluid and electrolyte homeostasis. In a collaborative project (Schweda et al. submitted), we show that the cardiac hormone "Brain Natriuretic Peptide", BNP (measured as the prohormone NT-pro-BNP), but not Atrial Natriuretic Peptide (ANP), could play an important role in this adaptation. Plasma [NT-proBNP] rapidly increases 6-fold in human kidney donors. The figure shows single kidney GFR (left) and plasma NT-proBNP (right) before total unilateral nephrectomy (UNx) and 4 days after in family kidney donors. In animal experiments, BNP infusion to mice increases GFR and RBF and targeted deletion of the receptor for BNP (GC-A) abolished these effects. BNP relaxed microdissected intrarenal human arteries isolated in our center. For termination of action, BNP depends to a large degree on renal excretion and thus our data could suggest an "automatic", built-in protective mechanism when renal function displays an acute decline. In fact, its clinical utility as a biomarker in cardiology for ventricular function/load is discussed in relation to its dependence on renal function for excretion. Thus renal dysfunction is a cause for elevated BNP in the absence of left ventricular dysfunction (7) It is clear that 1) NT-proBNP changes parallel to BNP, and 2) and they are equally dependent on renal function for their clearance (8). Degradation of peptides occur enzymatically and, of note, there is a beneficial effect of Dipeptidyl peptidase 4 (DPP4) inhibitors on kidney function during ischemic injury of kidney (9). Since BNP signals through a series of catalytic receptors with guanylyl cyclase activity and cyclic guanidine monophosphate (cGMP) formation, it is highly interesting that administration of phosphodiesterase-5 (PDE-5) inhibitor sildenafil improved immediate renal function in an kidney autotransplant pig model and in a warm ischemia-reperfusion pig model (10,11). Moreover, mice deficient in the receptor for ANP and BNP (GC-A) display hypertension. It is therefore likely that BNP increases acutely in the immediate post-nephrectomy phase which promotes glomerular filtration in remaining nephrons and contributes to maintain low blood pressure (12). There is a paucity of direct examinations of the mechanistic relationship between renal function and plasma BNP. This is now possible in a setting with acute surgical removal of defined renal mass. We aim to characterize acute and longitudinal changes in BNP (NT-proBNP) in patients with e.g partial nephrectomy and other "nephron-sparing" interventions and compare them to total nephrectomy patients with respect to correlation to GFR and prediction of long-term renal function.

Aim of the Study The overall aims are to preserve and protect remaining kidney function and improve the long-term renal outcome of renal surgical intervention with renal mass reduction.

Objective The project aim is to investigate the functional response and predictive significance of Brain Natriuretic Peptide (NT-proBNP) for renal function and blood pressure level after renal surgical intervention and in particular, to focus on the changes after partial nephrectomy compared to total nephrectomy.

Specific Hypotheses

1. The early plasma (5 days) [NT-proBNP] response predicts long-term total renal function and function of the remaining kidney (primary effect)
2. Plasma [NT-proBNP] increases acutely after partial nephrectomy and the change reflects the renal mass reduction
3. Chronic blood pressure change is inversely related to plasma [BNP] Design: The study is designed as an observational, longitudinal study where plasma [NT-proBNP], renal function and blood pressure is followed in patients undergoing partial or total nephrectomy ("nephron sparing surgery") and relate this to plasma BNP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suspected to have renal tumors by CT/Ultrasonic-scanning and eligible for intervention.
2. Healthy kidney donors scheduled for donation
3. Patients aged between 25 and 80 years
4. Patients can read and understand Danish

Exclusion Criteria:

1. Severe hypertension or congestive heart failure in New York Heart Association (NyHA) classes III-IV.
2. Renal insufficiency with glomerular filtration rate (eGFR) <50%
3. Failure to comply

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is designed as an observational, longitudinal study where plasma [NT-proBNP], renal function and blood pressure is followed in patients undergoing partial or total nephrectomy ("nephron sparing surgery") and relate this to plasma BNP.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
NT-proBNP | 5 days

SECONDARY OUTCOMES:
Partial nephrectomy_proBNP | 5 days
Chronic blood pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nessn Azawi, M.D., Study Chair — Roskilde University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Janzen NK, Kim HL, Figlin RA, Belldegrun AS. Surveillance after radical or partial nephrectomy for localized renal cell carcinoma and management of recurrent disease. Urol Clin North Am. 2003 Nov;30(4):843-52. doi: 10.1016/s0094-0143(03)00056-9. PMID 14680319
- [Result] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Result] Patel N, Sullivan M, Cranston D. Re: nephrectomy induced chronic renal insufficiency is associated with increased risk of cardiovascular death and death from any cause in patients with localized cT1b renal masses: C. J. Weight, B. T. Larson, A. F. Fergany, T. Gao, B. R. Lane, S. C. Campbell, J. H. Kaouk, E. A. Klein and A. C. Novick J Urol 2010; 183: 1317-1323. J Urol. 2010 Nov;184(5):2213-4; author reply 2214. doi: 10.1016/j.juro.2010.06.127. Epub 2010 Sep 22. No abstract available. PMID 20864134
- [Result] Becker F, Van Poppel H, Hakenberg OW, Stief C, Gill I, Guazzoni G, Montorsi F, Russo P, Stockle M. Assessing the impact of ischaemia time during partial nephrectomy. Eur Urol. 2009 Oct;56(4):625-34. doi: 10.1016/j.eururo.2009.07.016. Epub 2009 Jul 28. PMID 19656615
- [Result] Gill IS, Kavoussi LR, Lane BR, Blute ML, Babineau D, Colombo JR Jr, Frank I, Permpongkosol S, Weight CJ, Kaouk JH, Kattan MW, Novick AC. Comparison of 1,800 laparoscopic and open partial nephrectomies for single renal tumors. J Urol. 2007 Jul;178(1):41-6. doi: 10.1016/j.juro.2007.03.038. Epub 2007 May 11. PMID 17574056
- [Result] Azawi NH, Christensen T. Promising early results after hand-assisted laparoscopic partial nephrectomy in carefully selected patients. Dan Med J. 2012 Oct;59(10):A4520. PMID 23158896
- [Result] Luchner A, Hengstenberg C, Lowel H, Riegger GA, Schunkert H, Holmer S. Effect of compensated renal dysfunction on approved heart failure markers: direct comparison of brain natriuretic peptide (BNP) and N-terminal pro-BNP. Hypertension. 2005 Jul;46(1):118-23. doi: 10.1161/01.HYP.0000170140.36633.8f. Epub 2005 Jun 6. PMID 15939804